CLINICAL TRIAL: NCT04985604
Title: A Phase 2, Subprotocol of DAY101 Monotherapy for Patients With Recurrent, Progressive, or Refractory Solid Tumors With MAPK Pathway Aberrations
Brief Title: Tovorafenib (DAY101) Monotherapy for Patients With Melanoma and Other Solid Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Day One Biopharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAY101-102a; 2021-003768-29 (EudraCT Number)
Record Dates: First submitted 2021-06-23; First posted 2021-08-02 (Actual); Results first posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Melanoma; Solid Tumor; CRAF Gene Amplification; RAF1 Gene Amplification; BRAF Gene Fusion; BRAF Fusion; CRAF Gene Fusion; CRAF Fusion; RAF1 Gene Fusion; RAF1 Fusion; Thyroid Cancer, Papillary; Spitzoid Melanoma; Pilocytic Astrocytoma; Pilocytic Astrocytoma, Adult; Non Small Cell Lung Cancer; Non-Small Cell Adenocarcinoma; Colorectal Cancer; Pancreatic Acinar Carcinoma; Spitzoid Malignant Melanoma; Bladder Cancer; Bladder Urothelial Carcinoma; MAP Kinase Family Gene Mutation; RAF Mutation
Keywords: BRAF fusion; CRAF/RAF1 fusion; CRAF/RAF1 amplification
MeSH Terms: conditions — Melanoma; Thyroid Cancer, Papillary; Astrocytoma; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Pancreatic Neoplasms; Urinary Bladder Neoplasms | interventions — tovorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Melanoma Cohort (Experimental): Tovorafenib monotherapy
  Interventions: Drug: Tovorafenib
- Tissue Agnostic Cohort (Experimental): Tovorafenib monotherapy
  Interventions: Drug: Tovorafenib

INTERVENTIONS:
Drug: Tovorafenib — Tovorafenib tablet for oral use.
  Other Names: DAY101

SUMMARY:
This is a Phase 2, multi-center, open-label to evaluate the efficacy and safety of tovorafenib (DAY101) in participants ≥12 years of age with recurrent or progressive melanoma or solid tumors with BRAF fusion or CRAF/RAF1 fusions or amplification.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent by participants ≥ 12 years of age either a Consent or an Assent Form will be provided to the patient based on their capacity, local regulations, and guidelines.
* Participants must have a histologically confirmed diagnosis of melanoma or other solid tumor and a BRAF fusion, CRAF/RAF1 fusion, or CRAF/RAF1 amplifications obtained through a tumor or liquid biopsy as assessed by genomic sequencing, polymerase chain reaction (PCR), fluorescence in situ hybridization (FISH), or another clinically accepted molecular diagnostic method recognized by local laboratory or regulatory agency.
* Participants must have radiographically-recurrent or radiographically-progressive disease that is measurable using the appropriate tumor response criteria (e.g. RECIST version 1.1 or RANO).
* Archival tumor tissue (preferably less than 3 years old) or fresh tumor tissue for correlative studies is required
* If brain metastases are present, they must have been previously treated and be stable as assessed by radiographic imaging

Exclusion Criteria:

* Prior therapy of any RAS-, RAF-, MEK-, or ERK-directed inhibitor therapy
* Known presence of concurrent activating mutation
* Participants with current evidence or a history of central serous retinopathy (CSR), retinal vein occlusion (RVO)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-07-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (8):
  - The Angeles Clinic, Los Angeles, California
  - Hoag Health, Newport Beach, California
  - University of Colorado Hospital, Aurora, Colorado
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Community North Cancer Center, Indianapolis, Indiana
  - OHSU Knight Cancer Institute, Portland, Oregon
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
- Monash Medical Centre, Clayton, Victoria, Australia
- Antwerp University Hospital, Edegem, Belgium
- Canada (2):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
- Hopital de La Timone - APHM, Marseille, Bouches-du-Rhône, France
- South Korea (4):
  - Dong-A University Hospital, Busan
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (3):
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 11 centers that enrolled participants in 6 countries.
Pre-assignment Details: A total of 31 participants consented, of which 23 participants were enrolled into Melanoma and Tissue Agnostic cohorts. Remaining 8 participants were screen failures.
Groups:
- Melanoma Cohort: Adult participants (≥ 18 years) were administered Tovorafenib 600 mg orally (PO) once weekly (QW).
- Tissue Agnostic Cohort: Adult participants (≥ 18 years) were administered Tovorafenib 600 mg PO QW.
Period: Overall Study
Arm/Group | Melanoma Cohort | Tissue Agnostic Cohort
Started | 8 | 15
Completed | 4 | 8
Not Completed | 4 | 7
Not completed — Death | 4 | 6
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set comprised of all participants enrolled in the study who received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Melanoma Cohort | Tissue Agnostic Cohort | Total
Number analyzed (Participants) | 8 | 15 | 23
Age, Continuous [Median (Full Range); unit: Years] | 58.0 [26 to 71] | 45.0 [21 to 71] | 53.0 [21 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 4 | 8 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 7 | 14 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 10 | 13
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) by the Investigator
Description: ORR was defined as the percentage of participants with the best overall confirmed response of complete response (CR) or partial response (PR) according to the appropriate response assessment criteria including Response Evaluation Criteria in Solid Tumors (RECIST 1.1) or Response Assessment in Neuro-Oncology (RANO) for the disease setting as assessed by the Investigator. CR or PR was confirmed at a subsequent scan (>=4 weeks) if the criteria for each are met . The exact 95% confidence intervals (CIs) were calculated using Clopper-Pearson method.
Time Frame: Up to 23 months
Population: Efficacy Analysis Set comprises of all participants who received at least one dose of study drug and have measurable disease as determined by the Investigator at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Melanoma Cohort | Tissue Agnostic Cohort
Number analyzed (Participants) | 8 | 15
Percentage of participants | 50.0 [15.7 to 84.3] | 40.0 [16.3 to 67.7]

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An serious adverse event (SAE) is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or any other situation according to medical or scientific judgment. An AE is considered to be treatment-emergent if it has a start date/time on or after the first administration of study drug until 30 days after the last dose of study drug and before the start of subsequent therapy, whichever comes earlier. The distribution of AEs was analyzed by the type, frequency and severity for TEAEs.
Time Frame: Up to 23 months
Population: Safety Analysis Set comprises of all patients enrolled in the study who receive at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Melanoma Cohort | Tissue Agnostic Cohort
Number analyzed (Participants) | 8 | 15
Participants
  Any TEAE | 8 | 15
  TEAEs Related to Study Drug | 8 | 13
  Any serious TEAE | 2 | 8
  Serious TEAEs Related to Study Drug | 0 | 1
  TEAEs with Severity Grade 3 or Higher | 5 | 8
  TEAEs Related to Study Drug with Severity Grade 3 or Higher | 2 | 3
  TEAEs Leading to Death | 0 | 0
  TEAEs Related to Study Drug Leading to Death | 0 | 0
  TEAEs Leading to Study Drug Discontinuation | 1 | 0
  TEAEs Related to Study Drug Leading to Study Drug Discontinuation | 1 | 0

3. Secondary Outcome: Number of Participants With Worst Case Hematology Results by Maximum Grade Increase Post-baseline Relative to Baseline
Description: Blood samples were collected for the analysis of following hematology parameters: anemia, neutrophil count decreased and white blood cell decreased. Grade 1 (G1): mild; Grade 2 (G2): moderate; Grade 3 (G3): severe; Grade 4 (G4) life-threatening or disabling. Higher grade indicates greater severity and an increase in CTCAE grade was defined relative to the Baseline grade. Any worst-case post baseline increase to G2, G3, and G4 are presented. The laboratory parameters were graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.
Time Frame: Baseline and up to 23 months
Population: Safety Analysis Set comprises of all patients enrolled in the study who receive at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Melanoma Cohort | Tissue Agnostic Cohort
Number analyzed (Participants) | 8 | 15
Participants
  Anemia, Increased to Grade 2 | 3 | 5
  Anemia, Increased to Grade 3 | 2 | 2
  Anemia, Increased to Grade 4 | 0 | 0
  Neutrophil count decreased, Increased to Grade 2 | 0 | 2
  Neutrophil count decreased, Increased to Grade 3 | 0 | 1
  Neutrophil count decreased, Increased to Grade 4 | 0 | 0
  White blood cell decreased, Increased to Grade 2 | 0 | 2
  White blood cell decreased, Increased to Grade 3 | 0 | 0
  White blood cell decreased, Increased to Grade 4 | 0 | 0

4. Secondary Outcome: Number of Participants With Worst Case Chemistry Results by Maximum Grade Increase Post-baseline Relative to Baseline
Description: Blood samples were collected for the analysis of following chemistry parameters: creatine phosphokinase (CPK) increased, hypokalemia, hypoalbuminemia, hypercalcemia, hypocalcemia and hyponatremia. Grade 1 (G1): mild; Grade 2 (G2): moderate; Grade 3 (G3): severe; Grade 4 (G4) life-threatening or disabling. Higher grade indicates greater severity and an increase in CTCAE grade was defined relative to the Baseline grade. Any worst-case post baseline increase to G2, G3, and G4 are presented. The laboratory parameters were graded according to CTCAE version 5.
Time Frame: Baseline and up to 23 months
Population: Safety Analysis Set comprises of all patients enrolled in the study who receive at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Melanoma Cohort | Tissue Agnostic Cohort
Number analyzed (Participants) | 8 | 15
Participants
  CPK increased, Increased to Grade 2 | 2 | 4
  CPK increased, Increased to Grade 3 | 0 | 1
  CPK increased, Increased to Grade 4 | 1 | 0
  Hypoalbuminemia, Increased to Grade 2 | 1 | 2
  Hypoalbuminemia, Increased to Grade 3 | 0 | 0
  Hypoalbuminemia, Increased to Grade 4 | 0 | 0
  Hypokalemia, Increased to Grade 2 | 1 | 5
  Hypokalemia, Increased to Grade 3 | 0 | 1
  Hypokalemia, Increased to Grade 4 | 0 | 0
  Hyponatremia, Increased to Grade 2 | 1 | 1
  Hyponatremia, Increased to Grade 3 | 0 | 0
  Hyponatremia, Increased to Grade 4 | 0 | 0
  Hypercalcemia, Increased to Grade 2 | 0 | 0
  Hypercalcemia, Increased to Grade 3 | 0 | 1
  Hypercalcemia, Increased to Grade 4 | 0 | 0
  Hypocalcemia, Increased to Grade 2 | 0 | 1
  Hypocalcemia, Increased to Grade 3 | 0 | 0
  Hypocalcemia, Increased to Grade 4 | 0 | 0

5. Secondary Outcome: Duration of Response (DOR) in Participants With Best Overall Response
Description: Duration of response was defined as the interval from the date of the first documentation of tumor response (CR or PR) that was subsequently confirmed by investigator assessment to the date of first occurrence of radiographic disease progression based on RECIST 1.1 or RANO criteria or death due to any cause, whichever occurs earlier. DOR was estimated using Kaplan-Meier method.
Time Frame: Up to 23 months
Population: Participants in the Efficacy Analysis Set who have a confirmed response of CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Melanoma Cohort | Tissue Agnostic Cohort
Number analyzed (Participants) | 4 | 6
Months | 5.6 [3.0 to NA] — The upper bound of the 95% confidence interval was not estimable due to insufficient number of participants with events at the tail of the Kaplan-Meier curve. | 9.2 [3.5 to NA] — The upper bound of the 95% confidence interval was not estimable due to insufficient number of participants with events at the tail of the Kaplan-Meier curve.

6. Secondary Outcome: Duration of Progression Free Survival
Description: Progression free survival was defined as the interval from the date of the first dose to the first occurrence of radiographic disease progression based on RECIST 1.1 or RANO criteria or death due to any cause, whichever occurs earlier. Progression free survival was estimated using Kaplan-Meier method.
Time Frame: Up to 23 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Melanoma Cohort | Tissue Agnostic Cohort
Number analyzed (Participants) | 8 | 15
Months | 5.5 [1.8 to 12.5] | 5.5 [1.7 to NA] — The upper bound of the 95% confidence interval was not estimable due to insufficient number of participants with events at the tail of the Kaplan-Meier curve.

7. Secondary Outcome: Duration of Overall Survival
Description: Overall survival is defined as the interval from the date of the first dose until the recorded date of death due to any cause. Overall survival was estimated using Kaplan-Meier method.
Time Frame: Up to 23 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Melanoma Cohort | Tissue Agnostic Cohort
Number analyzed (Participants) | 8 | 15
Months | 18.9 [3.4 to NA] — The upper bound of the 95% confidence interval was not estimable due to insufficient number of participants with events at the tail of the Kaplan-Meier curve. | NA [5.5 to NA] — The median and upper bound of the 95% confidence interval was not estimable due to insufficient number of participants with events at the tail of the Kaplan-Meier curve.

8. Secondary Outcome: Time to Response
Description: Time to Response was defined in participants with best overall response of complete response or partial response as determined by Investigator. It is the interval from the date of the first dose to date of first documentation of tumor response that was subsequently confirmed by investigator assessment.
Time Frame: Up to 23 months
Population: Participants in the Efficacy Analysis Set who have a confirmed response of CR or PR were analyzed.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Melanoma Cohort | Tissue Agnostic Cohort
Number analyzed (Participants) | 4 | 6
Months | 1.76 [1.66 to 6.44] | 1.82 [1.77 to 1.87]

ADVERSE EVENTS:
Time Frame: Up to 23 months
Description: TEAE and serious TEAE were analyzed in Safety Analysis Set which comprised of all participants enrolled in the study who received at least one dose of tovorafenib.
Arm/Group | Melanoma Cohort | Tissue Agnostic Cohort
All-Cause Mortality (participants affected / at risk) | 4/8 | 6/15
Serious Adverse Events (participants affected / at risk) | 2/8 | 8/15
Other Adverse Events (participants affected / at risk) | 8/8 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Melanoma Cohort (N=8) | Tissue Agnostic Cohort (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Oedema (General disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Melanoma Cohort (N=8) | Tissue Agnostic Cohort (N=15)
Constipation (Gastrointestinal disorders) | 3 | 3
Vomiting (Gastrointestinal disorders) | 1 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Oral pain (Gastrointestinal disorders) | 0 | 2
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Face oedema (General disorders) | 3 | 2
Asthenia (General disorders) | 0 | 4
Fatigue (General disorders) | 4 | 0
Oedema (General disorders) | 1 | 2
Oedema peripheral (General disorders) | 0 | 3
Pyrexia (General disorders) | 0 | 3
Chills (General disorders) | 0 | 1
Gait disturbance (General disorders) | 0 | 1
Generalised oedema (General disorders) | 0 | 1
Influenza like illness (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 4
Rash (Skin and subcutaneous tissue disorders) | 3 | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 4
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 3
Acne (Skin and subcutaneous tissue disorders) | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 5 | 7
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 5
Alanine aminotransferase increased (Investigations) | 1 | 2
Weight decreased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 2
Blood bilirubin increased (Investigations) | 1 | 0
Blood calcium decreased (Investigations) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 1
Blood phosphorus decreased (Investigations) | 0 | 1
Tri-iodothyronine increased (Investigations) | 0 | 1
Troponin I increased (Investigations) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperchloraemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 2 | 1
Dizziness (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 0
Pyramidal tract syndrome (Nervous system disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 2
Vision blurred (Eye disorders) | 0 | 2
Blepharitis (Eye disorders) | 0 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 1
Eye disorder (Eye disorders) | 0 | 1
Eye pruritus (Eye disorders) | 0 | 1
Periorbital oedema (Eye disorders) | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 1
Vitreous detachment (Eye disorders) | 0 | 1
Vitreous floaters (Eye disorders) | 0 | 1
Influenza (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 2
COVID-19 (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Hordeolum (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Depression (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 1
Palpitations (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Embolism (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Lip injury (Injury, poisoning and procedural complications) | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (3):
  • Study Protocol: Sub-protocol DAY102-102a (2022-10-19): https://cdn.clinicaltrials.gov/large-docs/04/NCT04985604/Prot_000.pdf
  • Study Protocol: Umbrella (Master) Protocol- DAY102-102 (2022-10-13): https://cdn.clinicaltrials.gov/large-docs/04/NCT04985604/Prot_002.pdf
  • Statistical Analysis Plan (2024-04-12): https://cdn.clinicaltrials.gov/large-docs/04/NCT04985604/SAP_001.pdf